CLINICAL TRIAL: NCT03376360
Title: Optimization of 18F-choline PET/CT Acquisition in Prostate Cancer: Preliminary Results Concerning the Length of the Acquisition
Brief Title: Functional Medical Imaging Quantization in Prostate Cancer
Acronym: QUIP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: QUIP
Record Dates: First submitted 2017-11-24; First posted 2017-12-18 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; Fcholine; positron emission tomography; MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prostate cancer is the most common cancer in men over 50 years old and the third leading cause of cancer death. Because of the variety of prostate cancers, different treatments exist.

Several criteria guide this management in daily practice: PSA level; TNM stage (digital rectal examination, trans-rectal ultrasound and classical visual imaging) and pathological differentiation with the Gleason score, to which can be added other prognostic criteria: growth and doubling time of the serum PSA, number of positive biopsies and percentage of cancer lesions by biopsy.

Functional imaging by PET and MRI is increasingly used in daily clinical practice to characterize prostate cancer, either during initial discovery or during recurrence. In this context, it is the qualitative visual analysis that is mainly used. Quantitative image analysis could add new criteria to guide patient management.

Consequently, the objective of this study were:

* Optimization of 18F-choline PET/CT Acquisition in Prostate Cancer
* Comparison the quantitative parameters obtained by 18F-Choline PET / CT and both perfusion MRI and histological parameters.

ELIGIBILITY:
Inclusion Criteria:

Patients with prostate cancer histologically proven included in Brest University Hospital between 01/07/2012 and 01/10/2015 and underwent F-choline PET/CT and pelvic MRI Patient consent

Exclusion Criteria:

No lesion on dynamic acquisition on PET/CT and/or on pelvic MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer histologically proven included in Brest University Hospital between 01/07/2012 and 01/10/2015 and underwent F-choline PET/CT and pelvic MRI
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
correlation between Gleason score and dynamic parameters on PET and MRI | when anatomopathological report is available, an average of 3 months after the PET/CT
  study the potential correlation between dynamic parameters on PET and MRI

SECONDARY OUTCOMES:
reconstructions on 18F-choline PET | when all 18F-choline PET are performed, an average of 6 months
  determine the mean influx from each reconstruction which is the closest to the objective value
best "fitting" on PET and MRI | when all MRI are performed, an average of 6 months
  the Akaike Criteria Information was chose to choose the best fit
comparison between data (PSA, TNM stage, EFS and OS) | 01/05/2017
  comparison between data (PSA, TNM stage, EFS and OS)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France